CLINICAL TRIAL: NCT05332860
Title: Evaluation of Factors Affecting Extubation Times in Postoperative Congenital Cardiovascular Surgeries: A Randomized Prospective Study
Brief Title: Extubation Times in Postoperative Congenital Cardiovascular Surgeries
Status: Completed | Type: Observational
Sponsor: Bursa Yuksek Ihtisas Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Tugba Onur, Medical Doctor, Bursa Yuksek Ihtisas Training and Research Hospital
Other Study IDs: Bursa Education Hospital
Record Dates: First submitted 2022-03-22; First posted 2022-04-18 (Actual); Last update posted 2023-03-29 (Actual); Status verified 2023-03

CONDITIONS: Congenital Heart Disease
Keywords: Congenital heart disease; perioperative management; pediatric cardiac surgery; extubation
MeSH Terms: conditions — Heart Defects, Congenital

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Immediate Extubation or IE: patients were extubated in the operating room (OR) or in 6 hours after surgery
  Interventions: Procedure: Congenital Cardiovascular Surgery
- Early Extubation or EE: patients were extubated within 6-48 hours of admission to the ICU
  Interventions: Procedure: Congenital Cardiovascular Surgery
- Delayed Extubation or DE: patients were extubated sometime after 48 hours or not extubated
  Interventions: Procedure: Congenital Cardiovascular Surgery

INTERVENTIONS:
Procedure: Congenital Cardiovascular Surgery — Relationship between perioperative and postoperative hemodynamics, laboratory, oxygenation parameters and demographic data with extubation times in pediatric cardiac surgery cases taken in our hospital.

SUMMARY:
Background: Anesthesia management in pediatric cardiac surgeries focuses on reducing morbidity and mortality, early mobilization and discharge, using health resources sparingly and increasing the quality of life of patients. The duration of postoperative mechanical ventilation is one of the most important factors affecting the process after pediatric cardiac surgery. Besides the view that postoperative mechanical ventilation is safe, there are opposing views that it causes an increase in complications; It caused disagreements about extubation times. In our study, we aimed to investigate the factors affecting extubation times after pediatric cardiac surgery.

Methods: 72 ASA≥III pediatric patients undergoing cardiac surgery with cardiopulmonary bypass were included in our study. The patients were divided into 3 groups according to their extubation time. Those that were extubated in the operating room (OR) or in 6 hours after surgery (Immediate Extubation or IE), those that were extubated within 6-48 hours of admission to the ICU (Early Extubation or EE) and those that were extubated sometime after 48 hours or not extubated (Delayed Extubation or DE). Many variables of preoperative, peroperative and postoperative periods were recorded to see which factors correlated with extubation times.

DETAILED DESCRIPTION:
Children with critical congenital heart disease may need surgical or interventional procedures at some point in their lives.In pediatric cardiac anesthesia, it is important to reduce the need for postoperative mechanical ventilation in order to minimize morbidity, provide optimal vital functions, and reduce unnecessary use of health resources. Researchers aimed to examine the relationships of perioperative and postoperative hemodynamics, laboratory, oxygenation parameters and demographic data with extubation times in pediatric cardiac surgery cases taken in the hospital.

ELIGIBILITY:
Inclusion Criteria:

* elective or emergency patients
* aged 0-18 who are scheduled for congenital heart surgery

Exclusion Criteria:

-in patients who died during the operation

Ages: 1 Day to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: 72 patients
Sampling Method: Probability Sample
Enrollment: 72 (Actual)
Dates: Start 2020-05-01 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2021-02-15 (Actual)

PRIMARY OUTCOMES:
extubation times | 10 days after surgery
  postoperative mechanical ventilation times

SECONDARY OUTCOMES:
mortality | on 10 days
  mortality rates of groups

CONTACTS AND LOCATIONS:
Overall Officials: Tuğba T Onur, MD, Principal Investigator — Bursa Yuksek Ihtisas Training and Research Hospital; Ümran Ü Karaca, MD, Study Chair — Bursa Yuksek Ihtisas Training and Research Hospital; Anıl A Onur, MD, Study Chair — Bursa Yuksek Ihtisas Training and Research Hospital; Mesut M Engin, MD, Study Chair — Bursa Yuksek Ihtisas Training and Research Hospital; Asiye A Demirel, MD, Study Chair — Bursa Yuksek Ihtisas Training and Research Hospital; Halil Erkan HE Sayan, MD, Study Chair — Bursa Yuksek Ihtisas Training and Research Hospital; Şeyda Efsun ŞE Özgünay, MD, Study Chair — Bursa Yuksek Ihtisas Training and Research Hospital; Nermin N Kılıçarslan, MD, Study Chair — Bursa Yuksek Ihtisas Training and Research Hospital; Serkan S Seçici, MD, Study Chair — Bursa Yuksek Ihtisas Training and Research Hospital; Selimcan S Yırtımcı, MD, Study Chair — Bursa Yuksek Ihtisas Training and Research Hospital
Locations (1):
- Bursa Training and Research Hospital, Bursa, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided